CLINICAL TRIAL: NCT00077220
Title: Phase III Randomised Study Of Adjuvant Paclitaxel And Carboplatin (TAXOL-PARAPLATINE) With Concomittant Radiotherapy In Patients With Stage II or III Non-Metastatic Non-Small Cell Lung Cancer
Brief Title: Paclitaxel, Carboplatin, and Radiation Therapy With or Without Adjuvant Paclitaxel and Carboplatin in Treating Patients With Stage II or Stage III Unresectable Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000350015; FRE-GERCOR-B00-1; EU-20330
Record Dates: First submitted 2004-02-10; First posted 2004-02-11 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2007-05

CONDITIONS: Lung Cancer
Keywords: stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel; Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known whether giving chemotherapy together with radiation therapy is more effective with or without adjuvant chemotherapy in treating unresectable stage II or stage III non-small cell lung cancer.

PURPOSE: This randomized phase III trial is studying giving paclitaxel, carboplatin, and radiation therapy together with adjuvant paclitaxel and carboplatin to see how well it works compared to giving paclitaxel, carboplatin, and radiation therapy alone in treating patients with unresectable stage II or stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the progression-free survival of patients with stage II or III unresectable non-small cell lung cancer treated with paclitaxel, carboplatin, and radiotherapy with or without adjuvant paclitaxel and carboplatin.

Secondary

* Compare the objective response rate in patients treated with these regimens.
* Compare the overall survival of patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to radiotherapy regimen (conformational vs nonconformational).

Patients receive paclitaxel IV over 1 hour and carboplatin IV over 30 minutes once weekly for up to 6 weeks. Patients concurrently undergo radiotherapy 5 days a week for 7-7.5 weeks. Three weeks after completion of chemoradiotherapy, patients with stable or responding disease are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo routine follow-up.
* Arm II: Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for a maximum of 3 courses.

Patients are followed every 3 months for 2 years and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 390 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer

  * Stage II or III disease
  * Not amenable to surgery
* Measurable or evaluable disease
* No T4 apical localization
* Lesions able to be covered in a 60 Gy minimum volume of radiation
* No pleural effusion

PATIENT CHARACTERISTICS:

Age

* 18 to 79

Performance status

* ECOG 0-2

Life expectancy

* More than 3 months

Hematopoietic

* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3

Hepatic

* Bilirubin < 1.5 times upper limit of normal (ULN)

Renal

* Creatinine < 1.25 times ULN

Cardiovascular

* No unstable heart disease

Pulmonary

* No ventilation dysfunction that would preclude radiotherapy

Other

* No weight loss of 15% or more within the past 2 months
* No uncontrolled infection
* No other prior malignancy except curatively treated basal cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 6 months since prior neoadjuvant chemotherapy
* No prior adjuvant chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* No prior radiotherapy

Surgery

* Not specified

Other

* No other concurrent clinical trial participation

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-06

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Objective response rate
Overall survival
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Jean F. Morere, MD — Hopital Avicenne
Locations (68):
- France (68):
  - Centre Hospitalier d'Annecy, Annecy
  - Institut Sainte Catherine, Avignon
  - Hopital Duffaut, Avignon
  - Centre Hospitalier Bayeux, Bayeux
  - Centre Hospitalier de la Cote Basque, Bayonne
  - C.H.G. Beauvais, Beauvais
  - Hopital Avicenne, Bobigny
  - Clinique du Cedre, Bois-Guillaume
  - Hopital Saint Andre, Bordeaux
  - Clinique Tivoli, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Boucher
  - Polyclinique Du Parc Centre Maurice Tubiana, Caen
  - Hopital Louis Pasteur, Chartres
  - Centre d'Oncologie et de Radiotherapie de Chaumont le Bois, Chaumont
  - Centre Hospitalier Chaumont, Chaumont
  - Centre Hospitalier Chateaudun, Châteaudun
  - Hopital Louis Pasteur, Comar
  - Clinique des Cedres, Cornebarrieu
  - Centre d'Oncologie et de Radiotherapie du Parc, Dijon
  - Hopital Jean Monnet, Épinal
  - Centre Hospitalier D'Evreux, Évreux
  - Clinique Pasteur, Évreux
  - Clinique du Petit Colmouilins, Harfleur
  - Centre Mallet - Proux, Laval
  - C.H.G Laval, Laval
  - Centre Guillaume Le Conquerant, Le Havre
  - Centre Jean Bernard, Le Mans
  - C. H. Du Mans, Le Mans
  - Centre Hospitalier General, Le Mans
  - Hopital Robert Boulin, Libourne
  - Clinique de le Louviere, Lille
  - Clinique Chenieux, Limoges
  - Centre Hospitalier Robert Bisson, Lisieux
  - Medipole Gentilly Saint-Jacques, Maxéville
  - Hopital Notre-Dame de Bon Secours, Metz
  - Clinique du Pont de Chaume, Montauban
  - C.H. Du Havre, Montivilliers
  - Polyclinique Saint - Roch, Montpellier
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Clinique Clementville, Montpellier
  - Centre Hospitalier de Mulhouse, Mulhouse
  - Centre D'Oncologie De Gentilly, Nancy
  - Clinique De Valdegour, Nîmes
  - CHR D'Orleans - Hopital de la Source, Orléans
  - Hopital Saint-Louis, Paris
  - Hopital Tenon, Paris
  - C.H.G. De Pau, Pau
  - Maison Medicale Marzet, Pau
  - Clinique Saint - Pierre, Perpignan
  - Clinique les Bleuets, Reims
  - Groupe Medical St. Remy, Reims
  - Polyclinique De Courlancy, Reims
  - Centre Eugene Marquis, Rennes
  - Centre Frederic Joliot, Rouen
  - Centre Hospitalier de Saint - Brieuc, Saint-Brieuc
  - Clinique Armoricaine De Radiologie, Saint-Brieuc
  - Centre Rene Huguenin, Saint-Cloud
  - Centre Hospitalier De Saint Dizier, Saint-Dizier
  - Clinique Saint Vincent, Saint-Grégoire
  - Clinique de l'Union, Saint-Jean
  - Centre du Rouget, Sarcelles
  - C. H. De Saumur, Saumur
  - Clinique de l'Orangerie, Strasbourg
  - Polyclinique de L'Ormeau, Tarbes
  - Centre Hospitalier Regional Metz Thionville, Thionville
  - Centre Hospitalier de Valenciennes, Valenciennes
  - Clinique Medico Chirurgicale Teissier Groupe, Valenciennes
  - Centre Hospitalier De Vernon, Vernon